CLINICAL TRIAL: NCT00817154
Title: Individually Based Psychosocial Rehabilitation for Older People With SMI
Brief Title: Individually Based Psychosocial Rehabilitation for Older People With Serious Mental Illness (SMI)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: K23MH080021 (NIH)
Record Dates: First submitted 2009-01-05; First posted 2009-01-06 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-05

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Bipolar Disorder; Major Depression
Keywords: Older persons with SMI
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Bipolar Disorder; Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hopes-I (Experimental): The program progresses in three steps. First, participants receive a 10-week Basic Skills for Community Living course covering essential skills from each of the five modules to ensure that all participants establish basic competency in a core set of skills. Second, clinicians assess participants' functioning to identify skill areas that warrant additional improvement and engage participants in a shared decision making process to select skill areas to pursue in greater depth. Third, clinicians have weekly 60 minute sessions with participants in community settings for 7 months to provide training and to facilitate and support acquisition of core skills and rehabilitation goals.
  Interventions: Behavioral: HOPES-I

INTERVENTIONS:
Behavioral: HOPES-I — The program progresses in three steps. First, participants receive a 10-week Basic Skills for Community Living course covering essential skills from each of the five modules to ensure that all participants establish basic competency in a core set of skills. Second, clinicians assess participants' functioning to identify skill areas that warrant additional improvement and engage participants in a shared decision making process to select skill areas to pursue in greater depth. Third, clinicians have weekly 60 minute sessions with participants in community settings for 7 months to provide training and to facilitate and support acquisition of core skills and rehabilitation goals.

SUMMARY:
The major goal of this project is to adapt an existing group-based psychosocial program to enhance community functioning in older people with serious mental illness (SMI). The focus of the adaptation is designing and evaluating an individually based rehabilitative program for older people with SMI who either cannot or choose not to access a group program.

ELIGIBILITY:
Inclusion Criteria:

1. Age 50+;
2. ability to provide voluntary informed consent or assent, with formal consent by a legal guardian;
3. Axis I Disorder of schizophrenia, schizoaffective disorder, bipolar disorder, or major depression;
4. Functional impairment based on New Hampshire state eligibility criteria for services to people with SMI;
5. Enrollment in treatment for at least three months.

Exclusion Criteria:

1. residence in a nursing home or assisted living facility;
2. Terminal illness expected to result in death within one year or less;
3. Diagnosis of dementia, or significant cognitive impairment as indicated by a Mini Mental Status Evaluation (MMSE) score <24;
4. Current active substance abuse or dependence;
5. Past Participation in HOPES-G

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2009-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
To develop an individually based psychosocial rehabilitation program for older adults with SMI. The program will be specified in treatment manuals and will match relevant skills training modules to the functional needs and preferences of consumers. | baseline, 9 months and 12 months, 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Sarah I Pratt, Ph.D., Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (2):
- United States (2):
  - Riverbend Community Mental Health Center, Concord, New Hampshire
  - Community Council of Nashua, Nashua, New Hampshire